CLINICAL TRIAL: NCT02552745
Title: Sun Yat-sen University Cancer Center
Brief Title: Preventive Effects of Parecoxib on Postoperative Complications in Hepatocellular Carcinoma Patients Undergoing Hepatic Transcatheter Arterial Chemoembolization
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Department of Hepatobiliary Oncology, Sun Yat-sen University
Other Study IDs: B2012137
Record Dates: First submitted 2015-09-11; First posted 2015-09-17 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — parecoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: parecoxib sodium was administered postoperatively
  Interventions: Drug: parecoxib sodium
- control group: parecoxib sodium was not administered postoperatively

INTERVENTIONS:
Drug: parecoxib sodium — parecoxib sodium was administered postoperatively, when transcatheter arterial embolization finished.
  Groups: study group

SUMMARY:
This study is aiming to understand the effects of parecoxib on the postoperative complications of hepatocellular carcinoma (HCC) patients undergoing hepatic transcatheter arterial embolization (TACE). The investigators enrolled 242 patients who were diagnosed with HCC for the first time and who received hepatic TACE at the Cancer Prevention and Treatment Center of Sun Yat-sen University from October 2014 to March 2015 were prospectively enrolled. The patients were divided into study and control groups according to whether parecoxib sodium was administered postoperatively. Pain scores,body temperature, vomiting, and changes in liver function after surgery, as well as the length of the hospital stay, were recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with HCC according to the "primary liver cancer diagnosis and treatment practices" published by theMinistry of Health in 2011
2. A previous history of hepatitis B or positivity for hepatitis B surface antigen (HBsAg)
3. A Karnofsky Performance Status (KPS) score ≥70 points
4. Age between 18 and 65 years
5. Child-Pugh classA or B (class B patients had scores no greater than 7 points). In addition, the baseline laboratory tests had to meet the following criteria: white blood cells (WBCs) ≥1.5 × 109/L, platelets ≥50 × 109/L, hemoglobin ≥80 g/L, serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2 x the upper limit of normal (ULN), serum creatinine ≤ 1.5 x ULN, an international normalized ratio (INR)<1.5 or prothrombin time < the ULN + 4 seconds, albumin ≥30 g/L, and total bilirubin ≤34mmol/L

Exclusion Criteria:

1. Patients who had iodine allergies, severe heart and lung diseases, significant fever or pain, or continuous use of anti-inflammatory drugs within the past three months were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosed with HCC according to the "primary liver cancer diagnosis and treatment practices" published by the Ministry of Health in 2011 China.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pain scores | 3 days after TACE
  VAS pain scores recorded after TACE

SECONDARY OUTCOMES:
Body temperature | 3 Days after TACE
  The maximum daily temperature at each of the time points were recorded before TACE,two hours postoperative, and the first, second, and third postoperative days, respectively.
Liver function | 2 days after TACE
  Before and after TACE to compare
Hospital Stay | within 3 days after discharge